CLINICAL TRIAL: NCT06544759
Title: Confirmatory Factor Analysis (CFA) of a Questionnaire Used to Assess the Knowledge and Attitude of Medical Students Toward Organ Donation and Their Relationship With the Intent to Donate
Brief Title: Confirmatory Factor Analysis For A Questionnaire About Organ Donation
Status: Completed | Type: Observational
Sponsor: Rahmah Health Foundation (Other)
Collaborators: Rawalpindi Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: RHF-104-2024
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Tissue and Organ Procurement
Keywords: Organ Donation; Organ Graftings; Organ Procurement; Organ Procurement Systems; Organ Shortage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Aa educational Documentry — "The Gift of Life: Become an Organ Donor, Transform the Future!" is an informative and captivating documentary that delves into the world of organ transplantation and the powerful implications of organ donation. This documentary aims to dispel common misconceptions about organ donation and shares a heartwarming real-life story that highlights the life-saving potential of organ transplants. Through its comprehensive exploration of the subject and engaging storytelling, the documentary not only educates but also inspires profoundly. The documentary challenges preconceptions and aims to cultivate a culture of empathy, generosity, and life-saving commitment through its meticulous examination of the topic. The documentary serves as a powerful tool to raise awareness about the importance of organ donation and its potential to make a positive change in the world.

SUMMARY:
Purpose of the Study The study aims to understand how different messages can influence people's decisions to become organ donors. Researchers want to find out which types of messages are most effective in encouraging organ donation registration.

Who Can Take Part? Adults aged 18 and older who are eligible to register as organ donors can participate in this study.

How the Research Will Happen Participants will be shown different types of messages about organ donation. They will then be asked questions to see how the messages affect their willingness to register as organ donors. The study will compare the responses to determine which messages work best.

Benefits of the Study By identifying the most effective messages, this study aims to increase the number of registered organ donors. This can help save lives by making more organs available for transplantation.

DETAILED DESCRIPTION:
Background:

Organ donation is a vital component of modern healthcare, offering life-saving opportunities for patients with end-stage organ failure. Despite its importance, the number of registered organ donors remains insufficient to meet the demand for transplants. Previous research suggests that public perception and knowledge significantly influence the decision to register as organ donors. This study aims to assess the effectiveness of different messaging strategies on organ donation knowledge, attitudes, and intentions among medical students.

Objective:

The primary objective of this study is to evaluate the knowledge, attitudes, and intentions regarding organ donation among medical students. The study also aims to perform a Confirmatory Factor Analysis (CFA) on the questionnaire used to assess these factors.

Study Design:

This is a cross-sectional study with the following key elements:

Participants: Medical students aged 18 and older who are studying at [insert institution names or specify the institutions involved].

Intervention: Participants will receive different types of messages about organ donation. These messages will be crafted to appeal to various motivations and address common concerns about organ donation.

Data Collection: Participants will complete a questionnaire designed to evaluate their knowledge, attitudes, and intentions towards organ donation.

Procedure:

Recruitment: Participants will be recruited through announcements in medical schools, student organizations, and online platforms specific to medical students.

Message Delivery: Participants will be randomly assigned to receive one of several messages about organ donation through email, online platforms, or in-person sessions, depending on logistical feasibility.

Questionnaire Administration: After receiving the message, participants will complete a questionnaire that assesses their knowledge, attitudes, and intentions regarding organ donation. The questionnaire will be administered online or in-person.

Data Analysis: Confirmatory Factor Analysis (CFA) will be performed to validate the structure of the questionnaire. Statistical analyses will compare knowledge, attitudes, and intentions across different message groups.

Outcome Measures:

Primary Outcome: The primary outcome is the level of knowledge, attitudes, and intentions towards organ donation among medical students as measured by the questionnaire.

Secondary Outcomes: Secondary outcomes include the validation of the questionnaire structure through CFA and the identification of demographic factors that may influence the effectiveness of different messages.

Significance:

By assessing the effectiveness of various messaging strategies, this study aims to enhance educational approaches in medical schools regarding organ donation. Understanding medical students' perspectives on organ donation can help develop targeted educational interventions, potentially increasing the number of advocates for organ donation in the medical community.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate medical students in Pakistan who are proficient in English.

Exclusion Criteria:

* Participants who had previously taken part in organ donation awareness campaigns, undergone personal organ transplantation, or donated organs were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population consisted of undergraduate medical students from all years of the MBBS program in Pakistan. Participants were required to be proficient in English to ensure they could fully understand and respond to the study materials and questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Composite Score of Knowledge, Attitudes, and Intentions Towards Organ Donation | mmediately after message delivery (one-time assessment)
  The primary outcome measure is the composite score derived from the validated questionnaire, which assesses participants' knowledge, attitudes, and intentions regarding organ donation. This score will be calculated by summing responses to key items within the questionnaire that reflect these three domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Rahmah Health Foundation, Islamabad, Islamabad, Pakistan